CLINICAL TRIAL: NCT05112133
Title: Effect of Mulberry Leaf Extract on Glucose Response of a Test Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19.09 NRC
Record Dates: First submitted 2021-09-30; First posted 2021-11-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Post-prandial Glycemia
MeSH Terms: interventions — Morus alba; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Water administrated just before a meal
  Interventions: Dietary Supplement: Water
- Mulberry leaf extract before (Experimental): 250 mg of Mulberry leaf extract was administered before a standard meal
  Interventions: Dietary Supplement: Mulberry leaf extract
- Mulberry leaf extract during (Experimental): 250 mg of Mulberry leaf extract was administered during a standard meal
  Interventions: Dietary Supplement: Mulberry leaf extract

INTERVENTIONS:
Dietary Supplement: Mulberry leaf extract — Oral administration
  Arms: Mulberry leaf extract before; Mulberry leaf extract during
Dietary Supplement: Water — Oral administration
  Arms: Control

SUMMARY:
The aim of this study is to test the effects of Mulberry leaf extract on glucose response of a standardized complete meal when taken just before or when mixed with the meal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants
* Healthy status (based on anamnesis)
* Age between 18 and 45 years
* BMI between 20 and 29.9 kg/m2
* Ability to understand and sign an informed consent form

Exclusion Criteria:

* Pregnant or lactating women
* Major medical/surgical event in the last 3 months potentially interfering with study procedures and assessments
* Known food allergy and intolerance to test product
* Medically known cutaneous hypersensitivity to adhesives and plasters
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.

Smokers

Volunteer who cannot be expected to comply with the protocol

Subject having a hierarchical link with the research team members.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Post-prandial glucose | Hour 0 to hour 3 after standard meal consumption
  Incremental area under the curve

SECONDARY OUTCOMES:
C max glucose | Hour 0 to hour 3 after standard meal consumption
  Incremental C max
T max glucose | Hour 0 to hour 3 after standard meal consumption
  Incremental T max

CONTACTS AND LOCATIONS:
Locations (1):
- Nestlé Clinical Research Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided